CLINICAL TRIAL: NCT00629629
Title: Impacts of the 10 Steps for Healthy Feeding in Infants: a Randomized Field Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Marcia Regina Vitolo, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: vitolo2
Record Dates: First submitted 2008-03-05; First posted 2008-03-06 (Estimated); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Anemia; Breast Feeding, Exclusive; Overweight and Obesity
Keywords: Health Plan Implementation; Feeding and Eating Disorders of Childhood; Breastfeeding; Complementary feeding; Morbidity; Anemia; Public policy
MeSH Terms: conditions — Anemia; Breast Feeding; Overweight; Obesity; Feeding and Eating Disorders of Childhood | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Mothers in the intervention group received dietary advice based on Brazilian guidelines ["Ten steps for the healthy eating: Feeding guidelines for Brazilian children from birth to two years" ] during monthly home visits from 2 weeks to 6 months postpartum and then every 2 months thereafter until 1 y postpartum.
  Interventions: Behavioral: Dietary Advice
- Control (No Intervention): Mothers in the control group received routine medical assistance without any involvement of the research team. The study staff provided no materials to mothers on the Control Arm.

INTERVENTIONS:
Behavioral: Dietary Advice — Step 1 - Provide Exclusive breastfeeding up to 6 mo.
  Step 2- After 6 mo, gradually introduce complementary foods and continue breastfeeding up to 2 y or more.
  Step 3 - Complementary foods should be given 3 times a day (cereals, beans, fruits, and vegetables) if the child is breastfed, and 5 times a day if not.
  Step 4- Mealtimes must be adjusted to the children's cues of hunger and satiety.
  Step 5: Foods should gradually get thicker up to the time when the child is able to eat a family meal. Complementary foods should not be liquefied.
  Step 6: A large variety of healthy foods should be given daily to guarantee the intake of different nutrients.
  Step 7: Different fruits and vegetables should be offered daily. Step 8: Sugar, sweets, soft drinks, salty snacks, cookies, and processed and fried foods must be avoided.
  Step 9: Good hygiene practices in food preparation and handling.
  Step 10: Adequate feeding during child illness.
  Arms: Intervention

SUMMARY:
This study assesses the effectiveness of a nutrition advice programme - The ten steps for healthy feeding of children under two years old - on nutritional status, diet, and morbidity history of children. This is a randomized controlled trial in mostly socioeconomic deprived families (intervention=200; controls=300). Mothers of the intervention group received dietary counseling in the first year of life. Both groups received routine care by their paediatricians and research assessment at 6 and 12 months, 4 years, 8 years and 12 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants with birth weight ≥ 2.500 g and gestational age ≥ 37 weeks were considered eligible for the study.

Exclusion Criteria:

* HIV-positive mothers
* Congenital malformation
* Infants referred to intensive care unit
* Multiple pregnancy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2001-10; Primary Completion 2002-10 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Effectiveness of a nutrition advice programme in exclusive breastfeeding. | 1 year
  Group difference in months of esclusive breastfeeding
Effectiveness of a nutrition advice programme in dietary intake | 1 year
  Group differences in energy, fats, protein, carbohidrates and micronutrients intake
Effectiveness of a nutrition advice programme in dietary intake | 4 years
  Group differences in energy, fats, protein, carbohidrates and micronutrients intake
Effectiveness of a nutrition advice programme in dietary intake | 8 years
  Group differences in energy, fats, protein, carbohidrates and micronutrients intake
Effectiveness of a nutrition advice programme in dietary intake | 12 years
  Group differences in energy, fats, protein, carbohidrates and micronutrients intake

SECONDARY OUTCOMES:
Effectiveness of a nutrition advice programme in occurrence of diarrhea, respiratory problems, use of medication, dental caries,anemia and hospitalization. | 1 year
  Group differences in the % of children with each condition
Effectiveness of a nutrition advice programme in nutritional status | 1 year
  Group differences in the % of overweight and obese children.
Effectiveness of a nutrition advice programme in nutritional status | 4 years
  Group differences in the % of overweight and obese children.
Effectiveness of a nutrition advice programme in nutritional status | 8 Years
  Group differences in the % of overweight and obese children.
Effectiveness of a nutrition advice programme in nutritional status | 12 Years
  Group differences in the % of overweight and obese children.
Salty taste preferences | 12 years
  Evaluate the most preferred concentration of salt

CONTACTS AND LOCATIONS:
Overall Officials: Márcia R Vitolo, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre
Locations (1):
- Household, São Leopoldo, Rio Grande do Sul, Brazil

REFERENCES:
- [Result] Vitolo MR, Bortolini GA, Feldens CA, Drachler Mde L. [Impacts of the 10 Steps to Healthy Feeding in Infants: a randomized field trial]. Cad Saude Publica. 2005 Sep-Oct;21(5):1448-57. doi: 10.1590/s0102-311x2005000500018. Epub 2005 Sep 12. Portuguese. PMID 16158151
- [Result] Feldens CA, Vitolo MR, Drachler Mde L. A randomized trial of the effectiveness of home visits in preventing early childhood caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):215-23. doi: 10.1111/j.1600-0528.2006.00337.x. PMID 17518968
- [Derived] Valmorbida JL, Sangalli CN, Leffa PS, Baratto PS, Rauber F, Mennella JA, Vitolo MR. Sodium Intake Tracked from Infancy and Salt Taste Preference during Adolescence: Follow-up of a Randomized Controlled Field Trial in Brazil. Curr Dev Nutr. 2022 Dec 22;7(1):100011. doi: 10.1016/j.cdnut.2022.100011. eCollection 2023 Jan. PMID 37181123
- [Derived] Vitolo MR, da Costa Louzada ML, Rauber F, Campagnolo PD. Risk factors for high blood pressure in low income children aged 3-4 years. Eur J Pediatr. 2013 Aug;172(8):1097-103. doi: 10.1007/s00431-013-2012-9. Epub 2013 May 1. PMID 23636283
- [Derived] Louzada ML, Campagnolo PD, Rauber F, Vitolo MR. Long-term effectiveness of maternal dietary counseling in a low-income population: a randomized field trial. Pediatrics. 2012 Jun;129(6):e1477-84. doi: 10.1542/peds.2011-3063. Epub 2012 May 7. PMID 22566413
- [Derived] Bortolini GA, Vitolo MR. The impact of systematic dietary counseling during the first year of life on prevalence rates of anemia and iron deficiency at 12-16 months. J Pediatr (Rio J). 2012 Jan-Feb;88(1):33-9. doi: 10.2223/JPED.2156. Epub 2011 Dec 7. PMID 22159301
- [Derived] Vitolo MR, Rauber F, Campagnolo PD, Feldens CA, Hoffman DJ. Maternal dietary counseling in the first year of life is associated with a higher healthy eating index in childhood. J Nutr. 2010 Nov;140(11):2002-7. doi: 10.3945/jn.110.125211. Epub 2010 Sep 15. PMID 20844187
- [Derived] Feldens CA, Giugliani ER, Duncan BB, Drachler Mde L, Vitolo MR. Long-term effectiveness of a nutritional program in reducing early childhood caries: a randomized trial. Community Dent Oral Epidemiol. 2010 Aug;38(4):324-32. doi: 10.1111/j.1600-0528.2010.00540.x. Epub 2010 Apr 7. PMID 20406273